CLINICAL TRIAL: NCT06055075
Title: An Open-Label, Randomized Phase IB/II Study Evaluating Safety, Tolerability, and Clinical Activity of Forimtamig-Based Treatment Combinations in Participants With Relapsed or Refractory Multiple Myeloma
Brief Title: A Study Evaluating Safety, Tolerability, and Clinical Activity of Forimtamig-Based Treatment Combinations in Participants With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BP43437; 2023-503689-21-00 (EU CTIS Number)
Record Dates: First submitted 2023-09-20; First posted 2023-09-26 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Relapsed or Refractory Multiple Myeloma
MeSH Terms: conditions — Recurrence; Multiple Myeloma | interventions — carfilzomib; daratumumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Dose Exploration Phase: Forimtamig (Dose 1) + Carfilzomib (Experimental): Participants will receive Dose 1 of forimtamig, subcutaneous (SC) injection in combination with carfilzomib, intravenous (IV) infusion until disease progression.
  Interventions: Drug: Forimtamig; Drug: Carfilzomib
- Dose Exploration Phase: Forimtamig (Dose 2) + Carfilzomib (Experimental): Participants will receive Dose 2 of forimtamig, SC injection in combination with carfilzomib, IV infusion until disease progression.
  Interventions: Drug: Forimtamig; Drug: Carfilzomib
- Dose Exploration Phase: Forimtamig (Dose 3) + Carfilzomib (Experimental): Participants will receive Dose 3 of forimtamig, SC injection in combination with carfilzomib, IV infusion until disease progression.
  Interventions: Drug: Forimtamig; Drug: Carfilzomib
- Dose Exploration Phase: Forimtamig (Dose 1) + Daratumumab (Experimental): Participants will receive Dose 1 of forimtamig, SC injection in combination with daratumumab, SC injection until disease progression.
  Interventions: Drug: Forimtamig; Drug: Daratumumab
- Dose Exploration Phase: Forimtamig (Dose 2) + Daratumumab (Experimental): Participants will receive Dose 2 of forimtamig, SC injection in combination with daratumumab, SC injection until disease progression.
  Interventions: Drug: Forimtamig; Drug: Daratumumab
- Dose Exploration Phase: Forimtamig (Dose 3) + Daratumumab (Experimental): Participants will receive Dose 3 of forimtamig, SC injection in combination with daratumumab, SC injection until disease progression.
  Interventions: Drug: Forimtamig; Drug: Daratumumab
- Dose Expansion Phase: Forimtamig (Experimental): Participants will receive forimtamig, SC injection at a fixed dose determined during dose exploration phase until disease progression or completion of 12 months of treatment, whichever occurs first.
  Interventions: Drug: Forimtamig
- Dose Expansion Phase: Forimtamig + Carfilzomib (Experimental): Participants will receive forimtamig, SC injection at a fixed dose determined during dose exploration phase in combination with carfilzomib, IV infusion until disease progression.
  Interventions: Drug: Forimtamig; Drug: Carfilzomib
- Dose Expansion Phase: Forimtamig + Daratumumab (Experimental): Participants will receive forimtamig, SC injection at a fixed dose determined during dose exploration phase in combination with daratumumab, SC injection until disease progression.
  Interventions: Drug: Forimtamig; Drug: Daratumumab

INTERVENTIONS:
Drug: Forimtamig — Forimtamig will be administered SC at different doses during dose exploration phase. Forimtamig will be administered at a fixed dose determined during dose exploration phase in dose expansion phase.
Drug: Carfilzomib — Carfilzomib will be administered via IV infusion in combination with forimtamig.
  Arms: Dose Expansion Phase: Forimtamig + Carfilzomib; Dose Exploration Phase: Forimtamig (Dose 1) + Carfilzomib; Dose Exploration Phase: Forimtamig (Dose 2) + Carfilzomib; Dose Exploration Phase: Forimtamig (Dose 3) + Carfilzomib
Drug: Daratumumab — Daratumumab will be administered via SC injection in combination with forimtamig.
  Arms: Dose Expansion Phase: Forimtamig + Daratumumab; Dose Exploration Phase: Forimtamig (Dose 1) + Daratumumab; Dose Exploration Phase: Forimtamig (Dose 2) + Daratumumab; Dose Exploration Phase: Forimtamig (Dose 3) + Daratumumab

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and preliminary anti-tumor activity of forimtamig when administered alone or in combination with carfilzomib or daratumumab or other combination partners in participants with relapsed or refractory multiple myeloma (r/r MM). The study consists of two phases: a dose exploration phase and a dose-expansion phase.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Life expectancy of at least 12 weeks
* Documented diagnosis of MM according to the IMWG diagnostic criteria
* Evidence of progressive disease based on Investigator's determination of response by IMWG criteria on or after last dosing regimen
* Measurable disease
* AEs from prior anti-cancer therapy resolved to Grade ≤ 1,
* Adequate organ functions

Exclusion Criteria:

* Pregnant or breastfeeding or intending to become pregnant during the study or within 3 months after the last dose of study drug
* Plasma cell leukemia with circulating plasma cell count ≥ 5% or >500/microliter (µL)
* Participants with known amyloidosis
* Participants with myelodysplastic syndrome
* Prior treatment with monoclonal antibody (mAb) and antibody-drug conjugate within 4 weeks or 5 half-lives of the drug, whichever is shorter
* Prior anti-cancer therapy (chemotherapy, small molecule/tyrosine kinase inhibitors, radiotherapy) within 14 days prior to first forimtamig administration
* Prior solid organ transplantation
* Active auto-immune disease or flare within 6 months prior to start of study treatment
* Known or suspected chronic active Epstein-Barr virus (EBV) infection
* Hepatitis B virus (HBV) infection
* Acute or chronic hepatitis C virus (HCV) infection
* Known history of HIV seropositivity
* Live vaccine(s) within one month prior to start of the treatment
* Participants not fully vaccinated for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) as per local recommendations
* Previous refractoriness to carfilzomib
* Participants who discontinued prior carfilzomib treatment due to treatment-related toxicity
* Participants with known liver cirrhosis
* Participants eligible for allogeneic stem cell transplantation (SCT) or autologous SCT at the time of enrollment for Study BP43437 are excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2023-12-12 (Actual); Primary Completion 2025-07-08 (Actual); Study Completion 2025-07-08 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events (AEs) | Up to approximately 24 months
Objective Response Rate (ORR) as Determined by the Investigator per International Myeloma Working Group (IMWG) Criteria | Up to approximately 24 months
Complete Response (CR)/Stringent Complete Response (sCR) Rate as Determined by the Investigator per IMWG Criteria | Up to approximately 24 months
Rate of Very Good Partial Response (VGPR) or Better as Determined by the Investigator per IMWG Criteria | Up to approximately 24 months

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) as Determined by the Investigator per IMWG Criteria | Up to approximately 24 months
Duration of Response (DoR) for Participants who Achieve a Partial Response (PR) or Better as Determined by the Investigator per IMWG Criteria | Up to approximately 24 months
Time to First Response as Determined by the Investigator per IMWG Criteria | Up to approximately 24 months
Time to Best Response as Determined by the Investigator per IMWG Criteria | Up to approximately 24 months
Overall Survival (OS) as Determined by the Investigator per IMWG Criteria | Up to approximately 24 months
Serum Concentration of Forimtamig | Up to approximately 24 months
Percentage of Participants with Anti-Drug Antibodies (ADAs) to Forimtamig | Up to approximately 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (7):
- Australia (2):
  - Princess Alexandra Hospital Woolloongabba, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
- Hamilton Health Sciences, Hamilton, Ontario, Canada
- Istituto Clinico Humanitas, Rozzano, Lombardy, Italy
- New Zealand Clinical Research - Auckland, Auckland, New Zealand
- Seoul St Mary's Hospital, Seoul, South Korea
- Clinica Universitaria de Navarra, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing